CLINICAL TRIAL: NCT04464096
Title: Can Ankle and Foot Musculoskeletal Ultrasound Predict Fall Risk in Rheumatoid Arthritis Patients?
Brief Title: Can Musculoskeletal Ultrasound Predict Fall Risk in Rheumatoid Arthritis Patients?
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, safaa Mahran, Associate Proffesor, Assiut University
Other Study IDs: 17101098
Record Dates: First submitted 2020-06-18; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; foot problems; Fall risk; predictors
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non — non

SUMMARY:
Rheumatoid patients have higher fall risk than normal population. Several fall risk factors were studied. No previous study investigated the role of musculoskeletal ultrasound as a predictor of fall risk in rheumatoid arthritis.

DETAILED DESCRIPTION:
Adults with rheumatoid arthritis are exposed to higher risk of fracture. Risk factors included joint tenderness, fatigue, muscle weakness, impaired balance and disease activity.

Musculoskeletal ultrasound is a bed side radiographic tool that gained much attention in the last decade.It can detect stuctural chnges in the musculoskeletal system even before beeing detected by the x ray.

Nowadays, musculoskeletal ultrasound is a very useful tool in examining rheumatoid patients.

No previous study was done to investigate the role of musculoskeletal ultrasound as a predicting factor of fall risk in rheumatoid patients.

Predicting the fall risk in such disease could help setting preventing measures to prevent falls with its sequels.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Rheumatoid arthritis.

Exclusion Criteria:

* patients aged < 18 years
* Patients with lower limb disability preventing the participant from performing the mobility tests,
* Patients who were using antidepressants and sedatives.
* Patients with severe comorbidities, severe vision impairment, or hearing loss or neurological diseases that interferes with the mobility as stroke or neuropathy, were also excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with Rheumatoid arthritis .
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
range of motion | 1 week
  measured clinically as normal or restricted
muscle power | 1 week
  by manual testing with 5 grades where grade 5 means normal power
sensation | 1 week
  superficial sensation reported as intact or impaired
type of foot | 1 week
  using the wet test . three types of feet either normal, high arched or flat feet.
Tenitti balance assessment tool | 1 week
  The maximum total score is 28 points. In general, residents who score below 19 are at a high risk for falls
Berge Balance assessment | 1 week
  It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function A score of < 45 indicates individuals may be at greater risk of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
All data is treated confidentially.

REFERENCES:
- [Background] Stanmore EK, Oldham J, Skelton DA, O'Neill T, Pilling M, Campbell AJ, Todd C. Fall incidence and outcomes of falls in a prospective study of adults with rheumatoid arthritis. Arthritis Care Res (Hoboken). 2013 May;65(5):737-44. doi: 10.1002/acr.21892. PMID 23139011
- [Background] Hayashibara M, Hagino H, Katagiri H, Okano T, Okada J, Teshima R. Incidence and risk factors of falling in ambulatory patients with rheumatoid arthritis: a prospective 1-year study. Osteoporos Int. 2010 Nov;21(11):1825-33. doi: 10.1007/s00198-009-1150-4. Epub 2010 Jan 30. PMID 20119662
- [Background] Oswald AE, Pye SR, O'Neill TW, Bunn D, Gaffney K, Marshall T, Silman AJ, Symmons DP. Prevalence and associated factors for falls in women with established inflammatory polyarthritis. J Rheumatol. 2006 Apr;33(4):690-4. Epub 2006 Feb 15. PMID 16482644
- [Background] Armstrong C, Swarbrick CM, Pye SR, O'Neill TW. Occurrence and risk factors for falls in rheumatoid arthritis. Ann Rheum Dis. 2005 Nov;64(11):1602-4. doi: 10.1136/ard.2004.031195. Epub 2005 Apr 7. PMID 15817660